CLINICAL TRIAL: NCT06835036
Title: More Than Just p-Values: Minimal Clinically Important Difference for the Visual Analog Scale, Menstrual Symptom Questionnaire and Functional and Emotional Measure of Dysmenorrhea in Patients With Primary Dysmenorrhea
Brief Title: More Than Just p-Values: MCID for the VAS, MSQ and FEMD in Patients With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCID
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Primary Dysmenorrhea; Pain; Menstrual Discomfort
Keywords: Dysmenorrhea; Menstruation; Visual Analog Scale; Minimal Clinically Important Difference; ROC Curve
MeSH Terms: conditions — Pain; Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: In this prospective study, one treatment group was formed to receive exercise treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Treatment (Experimental): Each patient will receive a treatment protocol consisting of warm-up and functional exercises.
  Interventions: Other: Exercise Treatment

INTERVENTIONS:
Other: Exercise Treatment — In this study, a functional exercise programme will be performed 3 days a week for 8 weeks in three cycles as previously recommended. This programme consisted of a 5-minute warm-up and a 45-minute exercise phase.

SUMMARY:
The aim of this study is to determine the Minimal Clinically Important Difference (MCID) for the Visual Analog Scale (VAS), Menstrual Symptom Questionnaire (MSQ), and Functional and Emotional Measure of Dysmenorrhea (FEMD) in patients with primary dysmenorrhea (PwPD).

DETAILED DESCRIPTION:
100 PwPD will receive functional exercises three times a week for three menstrual cycles. Patients will be assessed on the most painful days of the first (baseline), second, and third menstrual cycles. The receiver operating characteristics (ROC) method and Gamma coefficient analysis will be applied to determine the responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the "No. 345-Primary Dysmenorrhea Consensus Guideline",
* Pain level of three or more according to VAS during activity (moderate to severe pain),
* Patients aged 18-35 years (when PD becomes more prevalent),
* Regular menstrual cycle with a duration of 28±7 days,
* Nulliparity.

Exclusion Criteria:

* Historical background of chronic urogenital infections or drug use,
* Pregnancy,
* Secondary dysmenorrhoea caused by gynaecological conditions such as endometriosis, adenomyosis and uterine fibroids.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with primary dysmenorrhea will be included.
Enrollment: 100 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (On the most painful day of the menstrual cycle before the intervention)
  Pain intensity in the lower abdomen, lower back and both thighs will be assessed using a 10 cm Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (excruciating pain). Pain levels were categorised as 0-2 (safe), 3-5 (acceptable) and 6-10 (risky).
Pain Intensity | After the 4-week intervention (On the most painful day of the first menstrual cycle after the start of the intervention)
  Pain intensity in the lower abdomen, lower back and both thighs will be assessed using a 10 cm Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (excruciating pain). Pain levels were categorised as 0-2 (safe), 3-5 (acceptable) and 6-10 (risky).
Pain Intensity | After the 8-week intervention (On the most painful day of the second menstrual cycle after the start of the intervention)
  Pain intensity in the lower abdomen, lower back and both thighs will be assessed using a 10 cm Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (excruciating pain). Pain levels were categorised as 0-2 (safe), 3-5 (acceptable) and 6-10 (risky).

SECONDARY OUTCOMES:
Menstrual Symptom Questionnaire (MSQ) | Baseline (On the most painful day of the menstrual cycle before the intervention)
  The Likert scale consists of 22 items, with responses rated on a 5-point range from 1 (never) to 5 (always). The scale includes three components: 'Negative Effects/Somatic Complaints' (items 1-13), 'Menstrual Pain Symptoms' (items 14-19), and 'Coping Methods' (items 20-22). The MSQ score is the mean value of all items in the scale. Increasing scores reflect more menstrual symptoms.
Menstrual Symptom Questionnaire (MSQ) | After the 4-week intervention (On the most painful day of the first menstrual cycle after the start of the intervention)
  The Likert scale consists of 22 items, with responses rated on a 5-point range from 1 (never) to 5 (always). The scale includes three components: 'Negative Effects/Somatic Complaints' (items 1-13), 'Menstrual Pain Symptoms' (items 14-19), and 'Coping Methods' (items 20-22). The MSQ score is the mean value of all items in the scale. Increasing scores reflect more menstrual symptoms.
Menstrual Symptom Questionnaire (MSQ) | After the 8-week intervention (On the most painful day of the second menstrual cycle after the start of the intervention)
  The Likert scale consists of 22 items, with responses rated on a 5-point range from 1 (never) to 5 (always). The scale includes three components: 'Negative Effects/Somatic Complaints' (items 1-13), 'Menstrual Pain Symptoms' (items 14-19), and 'Coping Methods' (items 20-22). The MSQ score is the mean value of all items in the scale. Increasing scores reflect more menstrual symptoms.
Functional and Emotional Measure of Dysmenorrhea (FEMD) | Baseline (On the most painful day of the menstrual cycle before the intervention)
  The FEMD is a 14-item measurement tool that evaluates the functional and emotional aspects of dysmenorrhea using a 5-point Likert-type scale. The total scores on this scale range from 14 to 70, with higher scores indicating a more significant functional and emotional impact of dysmenorrhea on an individual.
Functional and Emotional Measure of Dysmenorrhea (FEMD) | After the 4-week intervention (On the most painful day of the first menstrual cycle after the start of the intervention)
  The FEMD is a 14-item measurement tool that evaluates the functional and emotional aspects of dysmenorrhea using a 5-point Likert-type scale. The total scores on this scale range from 14 to 70, with higher scores indicating a more significant functional and emotional impact of dysmenorrhea on an individual.
Functional and Emotional Measure of Dysmenorrhea (FEMD) | After the 8-week intervention (On the most painful day of the second menstrual cycle after the start of the intervention)
  The FEMD is a 14-item measurement tool that evaluates the functional and emotional aspects of dysmenorrhea using a 5-point Likert-type scale. The total scores on this scale range from 14 to 70, with higher scores indicating a more significant functional and emotional impact of dysmenorrhea on an individual.
Global Rating Change (GRC) | After the 4-week intervention (On the most painful day of the first menstrual cycle after the start of the intervention)
  The GRC comprised seven responses, ranging from 1 to 7, indicating "very much better," "much better," "slightly better," "no change," "slightly worse," "much worse," and "very much worse," respectively.
Global Rating Change (GRC) | After the 8-week intervention (On the most painful day of the second menstrual cycle after the start of the intervention)
  The GRC comprised seven responses, ranging from 1 to 7, indicating "very much better," "much better," "slightly better," "no change," "slightly worse," "much worse," and "very much worse," respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Dr., Principal Investigator — Artvin Coruh University
Locations (1):
- Zeynep Yıldız Kızkın, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habibi N, Huang MS, Gan WY, Zulida R, Safavi SM. Prevalence of Primary Dysmenorrhea and Factors Associated with Its Intensity Among Undergraduate Students: A Cross-Sectional Study. Pain Manag Nurs. 2015 Dec;16(6):855-61. doi: 10.1016/j.pmn.2015.07.001. Epub 2015 Aug 29. PMID 26328887
- [Background] Guy M, Foucher C, Juhel C, Rigaudier F, Mayeux G, Levesque A. Transcutaneous electrical neurostimulation relieves primary dysmenorrhea: A randomized, double-blind clinical study versus placebo. Prog Urol. 2022 Jul;32(7):487-497. doi: 10.1016/j.purol.2022.01.005. Epub 2022 Mar 3. PMID 35249825
- [Background] Chesney MA, Tasto DL. The development of the menstrual symptom questionnaire. Behav Res Ther. 1975 Oct;13(4):237-44. doi: 10.1016/0005-7967(75)90028-5. No abstract available. PMID 1238078
- [Background] Li L, Huangfu L, Chai H, He W, Song H, Zou X, Wang W. Development of a functional and emotional measure of dysmenorrhea (FEMD) in Chinese university women. Health Care Women Int. 2012;33(2):97-108. doi: 10.1080/07399332.2011.603863. PMID 22242651
- [Background] Husted JA, Cook RJ, Farewell VT, Gladman DD. Methods for assessing responsiveness: a critical review and recommendations. J Clin Epidemiol. 2000 May;53(5):459-68. doi: 10.1016/s0895-4356(99)00206-1. PMID 10812317
- [Background] Burnett M, Lemyre M. No. 345-Primary Dysmenorrhea Consensus Guideline. J Obstet Gynaecol Can. 2017 Jul;39(7):585-595. doi: 10.1016/j.jogc.2016.12.023. PMID 28625286
- [Background] Myles PS. The pain visual analog scale: linear or nonlinear? Anesthesiology. 2004 Mar;100(3):744; author reply 745. doi: 10.1097/00000542-200403000-00042. No abstract available. PMID 15108996
- [Background] Yahaya Y, Ismail AH, Shamsuddin NH. Primary dysmenorrhoea among reproductive-age women at Kuala Selangor health clinic: Prevalence and factors associated. Med J Malaysia. 2022 Sep;77(5):569-575. PMID 36169068
- [Background] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122
- [Background] Kirmizigil B, Demiralp C. Effectiveness of functional exercises on pain and sleep quality in patients with primary dysmenorrhea: a randomized clinical trial. Arch Gynecol Obstet. 2020 Jul;302(1):153-163. doi: 10.1007/s00404-020-05579-2. Epub 2020 May 15. PMID 32415471
- [Background] Greco NJ, Anderson AF, Mann BJ, Cole BJ, Farr J, Nissen CW, Irrgang JJ. Responsiveness of the International Knee Documentation Committee Subjective Knee Form in comparison to the Western Ontario and McMaster Universities Osteoarthritis Index, modified Cincinnati Knee Rating System, and Short Form 36 in patients with focal articular cartilage defects. Am J Sports Med. 2010 May;38(5):891-902. doi: 10.1177/0363546509354163. Epub 2009 Dec 31. PMID 20044494
- [Background] Lehman LA, Velozo CA. Ability to detect change in patient function: responsiveness designs and methods of calculation. J Hand Ther. 2010 Oct-Dec;23(4):361-70; quiz 371. doi: 10.1016/j.jht.2010.05.003. Epub 2010 Jul 17. PMID 20638823